CLINICAL TRIAL: NCT05007561
Title: Understanding How Opioids Affect the Experiential and Neural Signatures of Social Experiences
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tristen Inagaki, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HS-2020-0188-SMT; R01DA052883 (NIH)
Record Dates: First submitted 2021-07-15; First posted 2021-08-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Naltrexone; Placebo
MeSH Terms: interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone (Experimental): 50mg naltrexone HCL once daily for seven days by mouth
  Interventions: Drug: Naltrexone Hydrochloride
- placebo (Placebo Comparator): sugar pill once daily for seven days by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — oral naltrexone
  Other Names: oral naltrexone; naltrexone pill; naltrexone; naltrexone oral tablet
  Arms: Naltrexone
Drug: Placebo — oral sugar pill
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The study is a randomized, placebo-controlled design with the opioid antagonist, oral naltrexone. Following random assignment, participants will take 50mg of naltrexone or placebo once a day for 7 days. On days 1 - 7, participants complete reports of their feelings of social connection and mood in order to assess more naturalistic feelings in response to opportunities for social connection outside of the laboratory setting. Additionally, at the end of each day, they complete a physical symptoms questionnaire. On the 7th day, participants will come to the SDSU MRI scanning facility to complete tasks designed to elicit feelings of social connection in the fMRI scanner. After the scan, feelings in response to the scanner tasks will be collected.

ELIGIBILITY:
Inclusion Criteria:

* good health
* English fluency
* willing to provide contact information for 4-6 close others
* willing to provide digital photographs of 2 close others
* own a smartphone

Exclusion Criteria:

* presence of medical devices, implants, or other metal objects in or on the body that cannot be removed
* tattooed eyeliner
* a body habitus prohibiting MRI scanning
* claustrophobia
* self-reported chronic mental or physical illness
* current and regular use of prescription medication
* previous history of having difficulty taking pills
* current use of opioid analgesics
* depressive symptoms above a 9 on Patient Health Questionnaire
* excessive alcohol use
* positive urine drug test
* body mass index (BMI) greater than 35
* pregnancy or plans to become pregnant in next 6 months
* positive urine pregnancy test

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Daily feelings of social connection via ecological momentary assessment | post-treatment, change across 7 days
  State feelings of social connection outside of the lab
Bold Oxygen-level Dependent (BOLD) Activations in Prespecified ROIs | Day 7, approximately 60 mins after taking study drug
  In the MRI scanner, participants read sentences written by people they know and people they do not know in a block design. In a second task they view images of people they know, those they do not know, and other emotional images. Brain activity will be measured as BOLD activity in response to stimuli from known (vs. unknown) people using functional magnetic resonance imaging (FMRI). Based on a priori hypotheses, brain activity will be masked to activity in structural regions-of- interest (ROIs) of the ventral striatum (VS), middle-insula (MI), anterior cingulate cortex (ACC) and ventromedial prefrontal cortex (VMPFC).
feelings in response to neuroimaging tasks | Day 7, approximately 150 minutes after taking study drug
  Feelings of social connection and general positive affect in response to the neuroimaging tasks will be reported on a scale of 1 (not at all) to 7 (very)

SECONDARY OUTCOMES:
physical symptoms via daily diary | end of day on days 1-7
  Physical symptoms previously associated with naltrexone will be assessed as well as the subjective experience of the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tristen Inagaki, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and resources from the current study will be deposited in the Open Science Framework (OSF) and OpenNEURO.org, in accordance with the NIH Data Sharing Policy. In addition, results will be posted on the ClinicalTrials.gov website within 1 year of the study's completion date.
Supporting Information: Analytic Code
Time Frame: After publication of the primary findings.
Access Criteria: Researchers in both private and public sector